CLINICAL TRIAL: NCT00574834
Title: Mechanisms of Reduced Ramipril on the Onset of Type 2 Diabetes Mellitis
Brief Title: Mechanisms of Ramipril Reduction in the Onset of Type 2 Diabetes
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00044872-Ramipril
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Ramipril; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ramipril (Active Comparator): Patients randomized to 6 months treatment of Ramipril.
  Interventions: Drug: Ramipril
- HCTZ (Active Comparator): PAtients randomized to 6 months treatment of HCTZ.
  Interventions: Drug: HCTZ-hydrochlorothiazide
- Ramipril+HCTZ (Active Comparator): Patients randomized to 6 months treatment of Ramipril+HCTZ.
  Interventions: Drug: Ramipril+HCTZ

INTERVENTIONS:
Drug: Ramipril — Ramipril 20 mg once daily for 6 months
  Other Names: Altace
  Arms: Ramipril
Drug: HCTZ-hydrochlorothiazide — HCTZ 25 mg once daily for 6 months
  Other Names: Brand Names: HydroDIURIL, Microzide
  Arms: HCTZ
Drug: Ramipril+HCTZ — Ramipril 20 mg and HCTZ 25 mg, both once daily for 6 months
  Other Names: Altace and HydroDIURIL, Microzide
  Arms: Ramipril+HCTZ

SUMMARY:
The study will be focused on determining the integrated in-vivo mechanisms responsible for Ramipril's effects on delaying type 2 diabetes and restoring normal (blood sugar levels) glycemia in patients with impaired glucose tolerance.

Hypothesis - Ramipril effects will delay the onset of type 2 diabetes and restore normal glycemia in patients with impaired glucose tolerance.

DETAILED DESCRIPTION:
Several studies have demonstrated that therapeutic agents used to reduce glucose levels and/or weight can delay the onset of type 2 diabetes. Intriguingly, angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB) also result in reduction in the onset of type 2 DM. The most striking effect was found with Ramipril in the HOPE study. The onset of new type 2 DM was reduced by 34% (p<0.001) as compared to placebo. Furthermore, the results of the DREAM trial demonstrate that Ramipril at a dose of 15 mg can significantly reverse impaired glucose tolerance. However, the mechanisms underlying Ramipril effects to delay type 2 diabetes are not known.

The proposal will be focused on determining the integrated in-vivo mechanisms responsible for Ramipril's effects on delaying type 2 DM and restoring normal glycemia in patients with impaired glucose tolerance.

The specific aims of the project are:

* to determine the effect of Ramipril on insulin resistance at the level of the liver and peripheral tissues,
* to determine the effect of Ramipril on endothelial function,
* to determine the effects of Ramipril on insulin secretion, and
* to determine the effects of Ramipril on substrate flux, lipolysis and inflammatory cytokines.

ELIGIBILITY:
Inclusion:

* 48 (24 male / 24 female) with impaired glucose tolerance.
* Impaired blood glucose values as outlined by the American Diabetes Association guideline. Fasting plasma glucose between 100 and 126 mg/dl or 2 hour post prandial glucose between 140 and 200 mg/dl
* BMI > 25 kgM2
* Age: 20-65 years
* Treated or Untreated hypertension defined as measurement of seated BP at screening visit of systolic BP 120 to 150 and/ or diastolic BP 80 to 100.

Exclusion:

* Patients receiving agents that can increase or lower blood glucose, i.e., metformin, thiazolidinediones, sulfonylureas, glitinides, acarbose, GLP-1 receptor agonists
* Untreated or treated while seated Systolic Blood pressure >150and/or Diastolic Blood pressure >100
* Taking hypertensive medications of HCTZ or ACE/ARB
* Allergy to HCTZ, heparin, nitroglycerin or lidocaine
* History of allergy or unacceptable side effects from ACE inhibitors
* Pregnancy or intent to become pregnant during the study
* Smoking
* Subject unable to give voluntary informed consent

Physical Exam Exclusion Criteria

* Clinically significant Cardiac Abnormalities (e.g. Heart Failure, Arrhythmia) from history or ECG in subjects > 40 years old
* Pneumonia
* Hepatic Failure/Jaundice
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit
* Fever greater than 38.0 C

Screening Laboratory Tests Exclusion Criteria according to protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, FRCP, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with pre-diabetes (metabolic syndrome) are recruited for a 6 month study intervention.
Period: Overall Study
Arm/Group | Ramipril | HCTZ | Ramipril+HCTZ
Started | 9 | 4 | 4
Completed | 9 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril | HCTZ | Ramipril+HCTZ | Total
Number analyzed (Participants) | 9 | 4 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 4 | 17
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (8.5) | 46 (9) | 41 (13) | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 6 | 1 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 6
  White | 6 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Changes in Insulin Sensitivity
Description: Measures of change in endogenous glucose production from baseline to final 30 minutes of clamp studies after 6 months of treatment.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Ramipril | HCTZ | Ramipril+HCTZ
Number analyzed (Participants) | 9 | 4 | 4
mg/kg/min | 0.98 (0.36) | 1.5 (0.23) | 1.2 (0.17)

ADVERSE EVENTS:
Arm/Group | Ramipril | HCTZ | Ramipril+HCTZ
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. No conclusions drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this trial were too preliminary to report. Trial was ended due to lack of funding to complete. No conclusions could be drawn from existing data.